CLINICAL TRIAL: NCT01059669
Title: A Multimodal Approach to Diagnose Patients With Chronic Pancreatitis
Brief Title: The Diagnosis of Chronic Pancreatitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Principal Investigator, Georg Gjorgji Dimcevski, MD, Haukeland University Hospital
Other Study IDs: REK nr 241.08
Record Dates: First submitted 2010-01-29; First posted 2010-02-01 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Pancreatitis
Keywords: Chronic pancreatitis; Pain; Exocrine insufficiency; Diabetes; Nutrition; Ultrasound
MeSH Terms: conditions — Pancreatitis, Chronic; Pain; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pankreatic juice Duodenal tissue Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients with suspected Chronic Pancreatitis
  Interventions: Other: diagnostic test
- Control group: Healthy controls
  Interventions: Other: diagnostic test

INTERVENTIONS:
Other: diagnostic test

SUMMARY:
To develop a new standardized multimodal diagnostic approach to CP considering:

WP 1: Fat in faeces and functional testing; the combination of tests has to be easy to practice, should take as little time as possible and discomfort for the patient has to be minimized WP 2: Advanced ultrasonography and imaging modalities. The focus is on validating standard parenchymal, contrast enhanced and functional ultrasound compared to a modern imaging standard. (CT, EUS, MRI)

To evaluate the reliability and feasibility of these novel methods in healthy volunteers; AND

To compare findings in known severe CP patients and different stages of pancreatic insufficiency in patients with CP.

DETAILED DESCRIPTION:
WP 1: Exocrine function testing

Aims:

Evaluating an endoscopic short test in patients with suspected pancreatic disease. Main focus on Chronic pancreatitis. (Collaborations to other patient groups in other protocols and to a group of healthy controls. )

Methods:

Secretintsimulated Endoscopic short test With duodenal sampling 30-45 minutes after secretin stimulation. Measurement of duodenal enzymes and duodenal bicarbonate concentration.

Inclusion:

Consecutive patients referred to a specialist outpatient clinic under suspicion of CP.

End Points:

Duodenal bicarbonate and enzyme concentrations. CP diagnosis by Layer/ Mayo score. Statistics: Simple comparishments of grpup means. Accuracy calculations by ROC curves. Sensitivity/ specificity calculations.

Sample size: Power and number of patients at baseline are calculated based on the following assumptions: The smallest difference between the pancreatic sufficient and the insufficient groups rejecting the null hypothesis are estimated to 25% regarding peak bicarbonate in EST. The worst case standard deviation is chosen 25%. Sample sizes of 14 patients in each group are expected to give the desired power of at least 0.80. Sample size: At least 15 patients in each group.

WP 2: Testing of Advanced ultrasound Methods

Aims:

Evaluate the diagnostic accuracy of transabdominal ultrasound (US) compared to CP diagnosis by Layer/ Mayo score, Endoscopic ultrasound (EUS), previous CT/ MRI examinations and exocrine pancreatic function.

Sample size:

Power and number of patients at baseline are calculated based on the following assumptions: The smallest difference between the pancreatic sufficient and the insufficient groups rejecting the null hypothesis are estimated to 35% regarding peak bicarbonate in traditional criteria counting. (average 4 criteria vs average 2 criteria) The worst case standard deviation is chosen 25%. Sample sizes of 14 patients in each group are expected to give the desired power of at least 0.80.

Sample size for interobserver variation analysis: Calculated by the principles of A Cantor(1). Assuming a relative error of 30% (Due to earlier observed large interobserver variations in these studies) , a clinical relevant kappa of 0.50 the estimated sample size must be above 44. We intended to include at least 60 patients with both US and EUS. In this setting kappa values below 0.4 must be interpreted with caution.

Hypothesis:

* US can demonstrate changes in CP
* US can diagnose CP with good accuracy.
* US can demonstrate minimal changes in CP
* US findings have good agreement compared to CP
* Changes by US correlate to severity by exocrine pancreatic function.

Inclusion criteria: : Consecutive adult patients (<16 years) referred to a specialized outpatient clinic with suspected chronic pancreatitis (CP) due to presenting symptoms or classical CP characteristics based on previous diagnostic imaging.

Exclusion criteria:

* Patients unable to give informed consent.
* Patients who had undergone extensive pancreatic surgery

In protocol exclusions pre-analysis:

* Subjects who did not fulfil the protocol for an adequate Mayo score
* Subjects with insufficient US visualization of the pancreas due to obesity, repeatedly overlying bowel air or other factors.

Methods:

* Collection of clinical data and previous CT/ MRI examinations from electrical patient journal. Nutritional screening with Height/ Weight/ BMI. Laboratory tests. Blood for DNA in Biobank,
* Exocrine function tests. Short endscopic secretintest/ Faecal Elastase
* Transabdominal Ultrasound: On inclusion and repeated 1-2 times within 3 months. Operators blinded to clinical data.

Registration of Rosemont criteria. Contrast enhanced ultrasound (CEUS) by Sonovue.

Endoscopic ultrasound: blinded to the results of the US. (Subjects offered conscious sedation with intravenous midazolam and pethidine or fentanyl hydrochloride during the test procedure) Pancreas Scan from head to tail. Parenchymal and ductal criteria registered.

Trial chronology:

1. In advance: Invited to participate. Written information in advance.
2. 1. Visit: Signed written consent. Anamnesis and nutritional score.

   o Ultrasound and EST
3. 2. Visit: Information of result.

   o Repeated ultrasound with registration of Rosemont criteria and CEUS
4. 3. Visit: EUS with Rosemont score.
5. 4. Visit: Follow up, Information of results. Plan further follow up and treatment.
6. Post analysis: Layer/ Mayo score. Rosemont/ traditional score of US and EUS

Endpoints:

CP diagnosis by Layer/ Mayo score Imaging scores: Traditional criteria count and Rosemont weighted score. Exocrine function results Endocrine function results Nutritional status results.

Statistical analysis:

Comparisons between groups are made using student t-tests or Mann-Whitney U-test as appropriate.

Accuracy data calculated from receiver operator curves (ROC). 5% level of statistical significance will be used. Interobserver variation for the separate criteria will be calculated as Cohens kappa.

Reliability for the ordinal data will be calculated as intraclass correlation coefficients (ICCs) in a random, two-way analysis. Data analyzed according to absolute agreement.

Agreement will be defined according to Landis and Koch: 0 = no agreement, 0 - 0.20 = slight agreement, 0.21 - 0.40 = fair agreement, 0.41 - 0.60 = moderate agreement, 0.61 - 0.80 = substantial agreement, and 0.81--1 = almost perfect agreement. A clinically relevant agreement usually requires a value >0.5.

Inclusion period: Starting from des 2009.

Reference List

1. Cantor A. Sample-Size calculations for Cohens Kappa. Psychological Methods 1996;1:150-153.

ELIGIBILITY:
Inclusion Criteria:

* The patients will be included from the Department of Medicine at Haukeland University Hospital in Norway. The Marseille-Rome diagnostic criteria will be used. Patients will be scored according to the Layer score. The symptoms should be unrelated to other systemic diseases.

Exclusion Criteria:

* Personality disturbances and alcohol consumption 24 hours prior to the study. Any other diseases and drugs associated with malabsorption; pregnancy or lactating women; heart disease or allergy against MR or ultrasound contrast agents.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient with suspected chronic pancreatitis age 18-67 years
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-08; Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Development of pancreatic insufficiency | 5 years
Peak enzyme Concentration IE | 5 Years

SECONDARY OUTCOMES:
development of diabetes | 5 years
Development of pain | 5 years
weight loss | 5 years
peak amylase | 5 Years

OTHER OUTCOMES:
lipase peak IE | 5 Years
Classical score US | 5 Years
Rosemont score US | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Georg Dimcevski, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway